CLINICAL TRIAL: NCT05191173
Title: Perioperative Three-dimensional Echocardiography in Cardioanesthesia.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: EchoRegistryCardiac
Record Dates: First submitted 2021-09-23; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Disease; Vascular Diseases
MeSH Terms: conditions — Heart Diseases; Vascular Diseases | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac Surgery — No intervention, just observation is performed.

SUMMARY:
The aim of this study is to investigate the significance of intraoperative echocardiography on the surgical course and association with patient outcome. Of particular interest is the three-dimensional assessment of cardiac and valvular function. The patient course from surgery to the time of hospital discharge will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery or surgery on the vessels near the heart

Exclusion Criteria:

* Pregnant patients
* Unfeasibility of intraoperative echocardiography in contraindications to transesophageal echocardiography: esophageal carcinoma, varices, diverticula, strictures, acute esophagitis, previous esophageal or gastric bleeding, symptomatic hiatal hernia.
* No written consent obtainable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mixed population of adult patients undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
In Hospital Mortality | up to 90 days
1-year Mortality | 1 year

SECONDARY OUTCOMES:
ICU Length of Stay | up to 90 days
Days on Mechanical Ventilation | up to 90 days
Days with Circulatory Support | up to 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No